CLINICAL TRIAL: NCT01577264
Title: Observational Study to Evaluate the Safety and Effectiveness of Cimzia in Rheumatoid Arthritis and Crohn's Disease Patients When Using a Comprehensive Program of Tuberculosis Screening and Monitoring
Brief Title: Certolizumab Pegol for the Treatment of Patients With Active Rheumatoid Arthritis (RA) and Crohn's Disease (CD)
Status: Terminated | Type: Observational
Why Stopped: Study is replaced by some Risk Manag. Activities covering the whole Russian Federation. Primary objectives could not be met due to critical missing information.
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: RA0091
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Rheumatoid Arthritis; Crohn's Disease
Keywords: Certolizumab Pegol; Cimzia
MeSH Terms: conditions — Arthritis, Rheumatoid; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cimzia treatment

SUMMARY:
This is an observational trial in Rheumatoid Arthritis and Crohn's Disease patients treated with Cimzia aiming to evaluate the risk and incidence of Tuberculosis.

DETAILED DESCRIPTION:
This is a prospective non interventional study. Patients enrolled in this study will receive Cimzia on prescription according to the instructions for use approved in Russia and within the frame of current standard clinical practices. The patient is evaluated at the Screening Visit for enrollment. A Baseline Visit is to be scheduled no more than 28 days after the Screening Visit. Subsequent evaluations are done routinely every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been prescribed Cimzia

Exclusion Criteria:

* Any contra-indication according to the Russian Summary of Product Characteristic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from previous UCB sponsored studies and all patients for whom the treating physician prescribed Cimzia.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2011-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Tuberculosis infection or reactivation during the study | From Baseline to Week 156 (Visit 7)
  The incidence of Tuberculosis (TB) infection or reactivation is assessed by routine TB diagnostic tests (Chest X-ray, skin test, Interferon-γ-release assays recognizing antigens representing 2 Mycobacterium tuberculosis proteins (preferably both blood and skin tests), ESAT-6 and CFP-10)

SECONDARY OUTCOMES:
Change from Baseline in Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) in Rheumatoid Arthritis (RA) patients at Week 26 | From Baseline to Week 26 (Visit 2)
  DAS28[ESR] is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity.
Change from Baseline in Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) in Rheumatoid Arthritis (RA) patients at Week 52 | From Baseline to Week 52 (Visit 3)
  DAS28[ESR] is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity.
Change from Baseline in Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) in Rheumatoid Arthritis (RA) patients at Week 78 | From Baseline to Week 78 (Visit 4)
  DAS28[ESR] is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity.
Change from Baseline in Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) in Rheumatoid Arthritis (RA) patients at Week 104 | From Baseline to Week 104 (Visit 5)
  DAS28[ESR] is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity.
Change from Baseline in Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) in Rheumatoid Arthritis (RA) patients at Week 130 | From Baseline to Week 130 (Visit 6)
  DAS28[ESR] is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity.
Change from Baseline in Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) in Rheumatoid Arthritis (RA) patients at Week 156 | From Baseline to Week 156 (Visit 7)
  DAS28[ESR] is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity.
Change from Baseline in Harvey Bradshaw Index (HBI) in Crohn's Disease patients (CD) at Week 26 | From Baseline to Week 26 (Visit 2)
  The HBI (Harvey and Bradshaw, 1980) will be calculated for all CD patients and is composed of 5 items:
  General well-being (0=Very well, 1=Slightly below Par, 2=Poor, 3=Very poor, 4=Terrible) Abdominal pain (0=None, 1=Mild, 2=Moderate, 3=Severe) Number of liquid stools per day Abdominal mass (0=None, 1=Dubious, 2=Definite, 3=Definite and tender) Complications (1 per item: Arthralgia, Uveitis, Erythema nodosum, Aphthous ulcers, Pyoderma gangrenosum, Anal fissure, New fistula, and Abscess)
Change from Baseline in Harvey Bradshaw Index (HBI) in Crohn's Disease patients (CD) at Week 52 | From Baseline to Week 52 (Visit 3)
  The HBI (Harvey and Bradshaw, 1980) will be calculated for all CD patients and is composed of 5 items:
  General well-being (0=Very well, 1=Slightly below Par, 2=Poor, 3=Very poor, 4=Terrible) Abdominal pain (0=None, 1=Mild, 2=Moderate, 3=Severe) Number of liquid stools per day Abdominal mass (0=None, 1=Dubious, 2=Definite, 3=Definite and tender) Complications (1 per item: Arthralgia, Uveitis, Erythema nodosum, Aphthous ulcers, Pyoderma gangrenosum, Anal fissure, New fistula, and Abscess)
Change from Baseline in Harvey Bradshaw Index (HBI) in Crohn's Disease patients (CD) at Week 78 | From Baseline to Week 78 (Visit 4)
  The HBI (Harvey and Bradshaw, 1980) will be calculated for all CD patients and is composed of 5 items:
  General well-being (0=Very well, 1=Slightly below Par, 2=Poor, 3=Very poor, 4=Terrible) Abdominal pain (0=None, 1=Mild, 2=Moderate, 3=Severe) Number of liquid stools per day Abdominal mass (0=None, 1=Dubious, 2=Definite, 3=Definite and tender) Complications (1 per item: Arthralgia, Uveitis, Erythema nodosum, Aphthous ulcers, Pyoderma gangrenosum, Anal fissure, New fistula, and Abscess)
Change from Baseline in Harvey Bradshaw Index (HBI) in Crohn's Disease patients (CD) at Week 104 | From Baseline to Week 104 (Visit 5)
  The HBI (Harvey and Bradshaw, 1980) will be calculated for all CD patients and is composed of 5 items:
  General well-being (0=Very well, 1=Slightly below Par, 2=Poor, 3=Very poor, 4=Terrible) Abdominal pain (0=None, 1=Mild, 2=Moderate, 3=Severe) Number of liquid stools per day Abdominal mass (0=None, 1=Dubious, 2=Definite, 3=Definite and tender) Complications (1 per item: Arthralgia, Uveitis, Erythema nodosum, Aphthous ulcers, Pyoderma gangrenosum, Anal fissure, New fistula, and Abscess)
Change from Baseline in Harvey Bradshaw Index (HBI) in Crohn's Disease patients (CD) at Week 130 | From Baseline to Week 130 (Visit 6)
  The HBI (Harvey and Bradshaw, 1980) will be calculated for all CD patients and is composed of 5 items:
  General well-being (0=Very well, 1=Slightly below Par, 2=Poor, 3=Very poor, 4=Terrible) Abdominal pain (0=None, 1=Mild, 2=Moderate, 3=Severe) Number of liquid stools per day Abdominal mass (0=None, 1=Dubious, 2=Definite, 3=Definite and tender) Complications (1 per item: Arthralgia, Uveitis, Erythema nodosum, Aphthous ulcers, Pyoderma gangrenosum, Anal fissure, New fistula, and Abscess)
Change from Baseline in Harvey Bradshaw Index (HBI) in Crohn's Disease patients (CD) at Week 156 | From Baseline to Week 156 (Visit 7)
  The HBI (Harvey and Bradshaw, 1980) will be calculated for all CD patients and is composed of 5 items:
  General well-being (0=Very well, 1=Slightly below Par, 2=Poor, 3=Very poor, 4=Terrible) Abdominal pain (0=None, 1=Mild, 2=Moderate, 3=Severe) Number of liquid stools per day Abdominal mass (0=None, 1=Dubious, 2=Definite, 3=Definite and tender) Complications (1 per item: Arthralgia, Uveitis, Erythema nodosum, Aphthous ulcers, Pyoderma gangrenosum, Anal fissure, New fistula, and Abscess)
Incidence of Adverse Events during the study | From Baseline to Week 156 (Visit 7)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (45):
- Russia (45):
  - 12, Kazan'
  - 16, Kazan'
  - 11, Moscow
  - 14, Moscow
  - 24, Moscow
  - 25, Moscow
  - 31, Moscow
  - 34, Moscow
  - 36, Moscow
  - 40, Moscow
  - 42, Moscow
  - 45, Moscow
  - 5, Moscow
  - 7, Moscow
  - 8, Moscow
  - 9, Moscow
  - 20, Orenburg
  - 21, Orenburg
  - 29, Orenburg
  - 43, Perm
  - 39, Petrozavodzk
  - 19, Saint Petersburg
  - 1, Saint Petersburg
  - 3, Saint Petersburg
  - 4, Saint Petersburg
  - 6, Saint Petersburg
  - 15, Samara
  - 18, Samara
  - 41, Samara
  - 33, Saratov
  - 17, Shakhty
  - 10, Taganrog
  - 26, Tolyatti
  - 22, Ufa
  - 27, Ufa
  - 32, Ufa
  - 35, Ufa
  - 37, Ufa
  - 38, Ufa
  - 55, Ufa
  - 30, Ulyanovsk
  - 23, Veliky Novgorod
  - 2, Yaroslavl
  - 13, Yekaterinburg
  - 28, Yekaterinburg